CLINICAL TRIAL: NCT00971919
Title: Prospective Cohort Study to Investigate Chronic Pain After Breast Cancer Surgery
Brief Title: Chronic Pain in Women Who Have Undergone Surgery for Stage I, Stage II, or Stage III Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aberdeen Royal Infirmary (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: EU-20926; CDR0000639659 (Registry Identifier: PDQ (Physician Data Query)); EU-20926
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-09

CONDITIONS: Breast Cancer; Pain; Perioperative/Postoperative Complications
Keywords: pain; perioperative/postoperative complications; breast cancer in situ; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Pain; Postoperative Complications; Breast Carcinoma In Situ | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Learning about chronic pain in women who have undergone surgery for breast cancer may help improve the quality of life for these patients and may help doctors plan the best treatment.

PURPOSE: This clinical trial is studying chronic pain in women who have undergone surgery for stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify which preoperative psychological risk factors, after controlling for demographic and clinical factors, are associated with chronic pain at 4 and 9 months after breast cancer surgery.
* Assess the incidence of chronic pain at 4 and 9 months after breast cancer surgery.
* Determine whether pain status at 4 and 9 months after breast cancer surgery is associated with changes in psychological well-being and health-related quality of life over time.

OUTLINE: This is a multicenter study.

Patients complete a preoperative pain questionnaire that includes the McGill Pain Questionnaire, a full body map, and the self-report Leeds Assessment of Neuropathic Symptoms and Signs scale. Only those patients with preoperative pain are asked to compete the full pain section of the questionnaire to assess location, severity, and type of pain. Acute postoperative pain during the first week after surgery is assessed using a visual analog scale (0-10). Patients then undergo telephone assessment of intensity and timing of acute pain 7 days after surgery. Subsequent postoperative pain assessments are conducted by mail using questionnaires at 4 and 9 months after surgery. Patients reporting chronic pain in the region of the surgical site are asked to complete the detailed pain section of the questionnaire.

Demographic variables, including age, education level, marital status, and body mass index, are recorded at baseline. Psychological (anxiety and exaggerated negative beliefs about pain) and quality-of-life outcomes are recorded at baseline and at 4 and 9 months postoperatively.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer or carcinoma in situ of the breast by core biopsy or fine needle aspiration

  * Newly diagnosed disease
  * Stage I-III disease
  * Resectable disease
* Being treated in the Aberdeen, Dundee, Perth, or Inverness Breast Unit

  * Planning to undergo primary surgical excision of the tumor (e.g., breast conservation surgery or mastectomy with or without axillary surgery [sentinel node biopsy, axillary sample, or axillary clearance])
  * Planning to undergo standard adjuvant therapy after surgery, including radiotherapy, chemotherapy, and/or hormonal therapy, as per existing standard protocols
* No detectable metastatic disease

PATIENT CHARACTERISTICS:

* Not pregnant
* Speaks English
* No history of mental illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Chronic pain at or near the surgical site persisting beyond the expected healing time as measured at 4 and 9 months after surgery
Identification of which psychological and quality of life variables, after controlling for baseline demographic, surgical, and other factors, are predictive of chronic pain at 4 and 9 months after surgery
Association between chronic pain status at 4 and 9 months after surgery and differential changes in quality-of-life outcomes since baseline

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bruce, MD, PhD, Principal Investigator — Aberdeen Royal Infirmary
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom